CLINICAL TRIAL: NCT03996629
Title: Impact of Clinical Pharmacist Interventions in Vitamin K Antagonists Management at One Teaching Hospital in Vietnam: A Randomized Controlled Trial
Brief Title: Impact of Clinical Pharmacist Interventions in Vitamin K Antagonists Management at One Teaching Hospital in Vietnam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Tien Hoang Tran, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UMCAM01
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Anticoagulation
Keywords: pharmacist-managed anticoagulation; warfarin; acenocoumarol
MeSH Terms: interventions — Patient Education as Topic; Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist-managed anticoagulation service (Experimental)
  Interventions: Other: Patient education and compliance
- Usual medical care (No Intervention)

INTERVENTIONS:
Other: Patient education and compliance — When the patient is enrolled in the intervention group, pharmacists provide medical education about the pathophysiology, medications, lifestyle, how to prevent, recognize and take care of bleeding events, etc. Establish a medical record for every follow-up examination and remind follow-ups by message, phone every month.
  Arms: Pharmacist-managed anticoagulation service

SUMMARY:
For decades, vitamin K antagonists are the main oral anticoagulants used for primary and secondary prevention of arterial and venous thromboembolic events. Both observational and randomized controlled trials have confirmed an outstanding outcome (the percentage of time in the therapeutic range-TTR, effectiveness and safety) in patients received anticoagulation management provided by pharmacists (AMPP) in comparing with usual physician care.

However, at present, pharmacist-managed anticoagulation services are still not popular in developing countries. In addition, there are few studies evaluating the patient outcomes with the AMPP model in Vietnam. Above all, it is important to explore whether AMPP is superior to other usual models in the improvement of effectiveness and safety.

DETAILED DESCRIPTION:
The study is a randomized controlled trial. Patients who will use VKA are prospectively divided into routine group and pharmacist intervention group.

For the intervention group, patients receive an intensive medical education from pharmacists in anticoagulation management service. Pharmacists regularly provide telephone and outpatient follow-up. At the end of the 12-month follow-up, the percentage of TTR and major bleeding events will be evaluated in both groups.

Clinical data is designed to be collected from 800 patients, 400 patients in each group. Data will be analyzed by SPSS 20.0 software. P < 0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients received a discharge prescription with VKA therapy from November 2018
* Patients agree to participate in the study
* Age 18 and older
* Duration of VKA therapy ≥12 months

Exclusion Criteria:

* Patients with cognitive impairment as diagnosed by physician
* Geographical and financial conditions do not allow patients to guarantee follow-up examination on schedule
* Patient has less than 3 INR test results after the first day participating in the study
* Cannot contact patient by phone call or face-to-face communication after the first day participating in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Time in the therapeutic range (TTR) | 12 months
  The time in the therapeutic range (TTR) has been used as a measure of warfarin therapy quality. The percentage of TTR is the percentage of the number of patient's INR achieved therapeutic range on the total number of patient's INR test in the 12-month follow-up of each patient.
Bleeding events | 12 months
  Major bleeding is considered to be those events that resulted in death or the need for acute medical or surgical intervention, also as defined by previously described criteria. Minor bleeding includes increased bruising on the skin and other bleeding episodes not meeting the criteria for major bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Trang Dang, PhD, Study Chair — University Medical Center Ho Chi Minh City
Locations (1):
- University Medical Center Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No